CLINICAL TRIAL: NCT02162134
Title: Does Sugared or Sugar Free Chewing Gum Reduces Postoperative Ileus After Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benazir Bhutto Hospital, Rawalpindi (Other Government)
Responsible Party: Principal Investigator, Dr.Fazal hussain Shah, General Surgery Resident, Benazir Bhutto Hospital, Rawalpindi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BenazirBH
Record Dates: First submitted 2014-06-06; First posted 2014-06-12 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Postoperative Ileus.
Keywords: cholecystectomy; laparoscopic; postoperative; ileus; chewing gum
MeSH Terms: conditions — Ileus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- no chewing gum. (Other): the no chewing gum group was control and receive no chewing gum postoperatively. While they received all other medications like anesthesia, antibiotics etc
  Interventions: Drug: Tab. Midazolam 7.5 mg; Drug: Inj. Midazolam 0.7mg/kg 45 min before surgery; Drug: Inj. Propofol 2.5mg/kg; Drug: Inj. Atracurium 0.5 mg/kg; Drug: Sevoflurane 2.5 vol %; Drug: Inj. Cefuroxime 1.5 g IV; Drug: Inj. Ketorolac 30 mg IV; Drug: Inj. Zantac 50mg IV
- sugar free chewing gum (Experimental): sugar free chewing was given to patients 4 hours after surgery then continue it 8 hourly (20 to 25 minutes each time) until oral feeding is started.
  Interventions: Other: sugared chewing gum; Drug: Tab. Midazolam 7.5 mg; Drug: Inj. Midazolam 0.7mg/kg 45 min before surgery; Drug: Inj. Propofol 2.5mg/kg; Drug: Inj. Atracurium 0.5 mg/kg; Drug: Sevoflurane 2.5 vol %; Drug: Inj. Cefuroxime 1.5 g IV; Drug: Inj. Ketorolac 30 mg IV; Drug: Inj. Zantac 50mg IV
- sugared chewing gum (Experimental): sugared chewing gum will be given 4 hours after surgery then continue it 8 hourly (20 to 25 minutes each time) until oral feeding is started
  Interventions: Other: sugar free chewing gum; Drug: Tab. Midazolam 7.5 mg; Drug: Inj. Midazolam 0.7mg/kg 45 min before surgery; Drug: Inj. Propofol 2.5mg/kg; Drug: Inj. Atracurium 0.5 mg/kg; Drug: Sevoflurane 2.5 vol %; Drug: Inj. Cefuroxime 1.5 g IV; Drug: Inj. Ketorolac 30 mg IV; Drug: Inj. Zantac 50mg IV

INTERVENTIONS:
Other: sugar free chewing gum — Sugar free chewing gum (orbit) was given to patients. They were asked to chew it 4 hours after surgery and continue to chew it 8 hourly for 20 to 25 min each time until oral feeding was started.
  Other Names: Orbit
  Arms: sugared chewing gum
Other: sugared chewing gum — Sugared chewing gum (singsong bubble gum) was given to patients. They were asked to chew it 4 hours after surgery and continue to chew it 8 hourly for 20 to 25 min each time until oral feeding was started.
  Other Names: Dingdong bubble gum.
  Arms: sugar free chewing gum
Drug: Tab. Midazolam 7.5 mg — Tab. Midazolam 7.5 mg will be given to all patients at night before surgery.
Drug: Inj. Midazolam 0.7mg/kg 45 min before surgery — Inj . Midazolam 0.7 mg/kg given as premedication.
Drug: Inj. Propofol 2.5mg/kg — It was given to induce anesthesia after 3 min of pre oxygenation.
Drug: Inj. Atracurium 0.5 mg/kg — It was given to induce muscle relaxation during anesthesia.
Drug: Sevoflurane 2.5 vol % — It was given to maintain anesthesia during surgery alongwith oxygen in air mixture
Drug: Inj. Cefuroxime 1.5 g IV — It was given as prophylactic antibiotic. 2 doses given. 1st 30-60 min before surgery. 2nd 6 hours after surgery
Drug: Inj. Ketorolac 30 mg IV — 3 doses for analgesia. 1st immediate postoperative, 2nd at 8 hours postoperative and 3 rd at 16 hours postoperative period.
Drug: Inj. Zantac 50mg IV — 2 doses. 1st at immediate postoperative and 2nd 12 hours after surgery

SUMMARY:
Laparoscopic cholecystectomy is now very common procedure to remove the gall bladder from abdomen. After this procedure many patients suffer from the non functioning of intestine and stomach which is very common after any abdominal surgery. Many efforts tried to reduce this non functioning period or postoperative ileus but non of them was superior later on. The investigators want to evaluate the role of chewing gum for reducing postoperative ileus. The investigators hypothesis is that Chewing gum after laparoscopic cholecystectomy reduces postoperative ileus and sugared preparations are more effective to reduce it.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy is considered now the gold standard for gall stone disease. Postoperative ileus after any abdominal surgery is common complication, it is considered as physiological response and is the main cause of postoperative abdominal pain, discomfort and increased duration of hospital stay. Postoperative ileus (POI) may last up to 5 days after uncomplicated abdominal surgery. Activity of small intestine returns within 24 hours while stomach and large intestine take up to 36 and 72 hours to regain motility.3 The use of early feeding, medications like cisapride etc. have been used to reduced POI but none of them has been significantly useful on further research work.

Gum chewing after abdominal surgery reduces the duration of POI, pain and discomfort. Gum chewing also reduces halitosis, dental caries, elevates mood and reduces stress which are additional benefits. Many studies proved that the chewing gum has only placebo effect after surgery in adults and children. Sugar-free chewing gum has been focused mainly in studies. Perioperative role of glucose intake has shown many benefits like reducing insulin resistance.

In this study the investigators wanted to evaluate the role of chewing gum in reducing POI in laparoscopic cholecystectomy and further exploration to see the whether which chewing gum is more beneficial, sugar-free or sugared. If the study proves the beneficial effect of chewing gum then the investigators can have better management of patients postoperatively by sugared chewing gum which is readily available and inexpensive.

After meeting inclusion and exclusion criteria, All patients were given Tab. Midazolam 7.5 mg PO at night before surgery and received same standard general anesthesia with endotracheal intubation. Inj. Midazolam IV 0.7 mg/kg was given 45 min before surgery as premedication. Anesthesia was induced by propofol (2.5 mg/kg) after 3 minutes of preoxygenation. Muscle relaxation was achieved by atracuium (0.5 mg/kg). Anesthesia was maintained with sevoflurane (2.5 vol %) and oxygen in air mixture (0.50 ratio). Ventilation was controlled mechanically and end tidal normocapnia was maintained by keeping pCO2 at 35-38 mmHg.

Following medications were given to patients during the process.

* Inj. Cefuroxime 1.5 gm. IV (2 doses, 1st dose 30-60 min before surgery and 2nd dose 6 hours after surgery)
* Inj. Ketorolac 30mg IV (3 doses total, 1st dose immediate postop, 2nd and 3rd at 8 and 16 hours after surgery respectively)
* Inj. Zantac 50 mg IV (2 doses total, 1st immediate postop and 2nd at 12 hours after surgery) All patients were operated by the consultant surgeons. Duration of surgery was noted. Patients were divided randomly into 3 groups equally; at the end each contained 30 patients each. Group A was the control group, group B received sugar-free chewing gum (Orbit) and group C received sugared chewing gum (Dingdong chewing gum from hilalcandy). Both B and C groups were asked to start chew gum 4 hours after surgery then continue it 8 hourly (20-25 minutes each time) until oral feeding was started. Onset of hunger, bowel movements, flatus passing and defecation were noted. Bowel movements were examined via stethoscope hourly after surgery. All patients received same standard postoperative care.

All the data was recorded on specially designed Performa. Statistical analysis: Data was analyzed using SPSS version 12. Mean and standard deviation were calculated for quantitative data like age, duration of surgery, time of onset of hunger, bowel movements, flatus passing and defecation. Frequency and percentages were calculated for qualitative data like gender. The results were finally analyzed and compared for the three groups using one way ANOVA. The data of any two groups (A versus B, A versus C, B versus C) was analyzed by independent sample t test. Pearson correlation was used to see the correlation between duration of surgery and bowel movements. A p value <0.05 was considered significant

ELIGIBILITY:
Inclusion Criteria

1. Patients undergoing elective laparoscopic cholecystectomy for gallstone disease.
2. Patients with age range of 25 to 55 years

Exclusion Criteria

1. H/O chronic illness like DM, IHD, CRF, CLD
2. Immunocompromised patients.
3. Previous history of any chemotherapy or radiotherapy, any history of repeated infections, pneumonia.
4. Patients with H/O concurrent intestinal illnesses like Tuberculosis, ulcerative colitis, Crohn's disease, acute or chronic diarrhea, constipation etc.
5. Previous hepatobilliary surgery.
6. H/O use of antispasmodics, or drugs affecting the intestinal motility within last 72 hours before and after surgery (tricyclic antidepressants, antipsychotics)
7. Patients who develop the postop complications like wound infection, intra-abdominal collections etc.
8. Complicated cholecystectomy in which laparoscopic cholecystectomy is converted to open cholecystectomy.
9. Cholecystectomy in which the biliary leakage was complication, either in the drain or later on detected via ultrasound

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2013-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
onset of hunger | 4 hours after surgery until patient feels first feeling of hunger. an expected average of 12 hours.
  the patients were asked when they felt first feeling of hunger. this time was noted in terms of hours after surgery.
onset of bowel movements | 4 hours after surgery until the bowel sounds are present. an expected average of 10 hours.
  the patients were examined by resident doctor hourly after surgery for presence of bowel sounds by a stethoscope. Additional all patient were asked when they felt first bowel sounds. the time at which the first bowel activity was present was noted in terms of hours after surgery.
onset of flatus passing | 4 hours after surgery until patient passes flatus. an expected average of 18 hours.
  the patients were asked when they passed first flatus. this time was noted in terms of hours after surgery.
onset of defecation | 4 hours after surgery until patient defecated. an expected average of 24 hours.
  the patients were asked when they passed stool first time after surgery. that time was noted in terms of hours after surgery.

SECONDARY OUTCOMES:
time of surgery | skin incision to skin closure time of surgery. an expected average of 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Fazal Hussain Shah, FCPS-I, Principal Investigator — Benazir Bhutto Hospital, Rawalpindi; Aurangzeb khan, FCPS, Study Chair — Benazir Bhutto Hospital, Rawalpindi; Muhammad Bilal Habshi, FCPS-I, Study Chair — Benazir Bhutto Hospital, Rawalpindi; Arslan Zahid, FCPS-I, Study Chair — Benazir Bhutto Hospital, Rawalpindi; Muhammad Zubair Saeed, FCPS-I, Study Chair — Benazir Bhutto Hospital, Rawalpindi
Locations (1):
- General Surgery Dept. Benazir Bhutto Hospital Rawalpindi, Rawalpindi, Punjab Province, Pakistan

REFERENCES:
- [Background] Gorski JP, Marks SC Jr, Cahill DR, Wise GE. Developmental changes in the extracellular matrix of the dental follicle during tooth eruption. Connect Tissue Res. 1988;18(3):175-90. doi: 10.3109/03008208809016806. PMID 3219849
- [Background] Lohrmann DK, Gold RS, Jubb WH. School health education: a foundation for school health programs. J Sch Health. 1987 Dec;57(10):420-5. doi: 10.1111/j.1746-1561.1987.tb03187.x. PMID 3326971
- [Background] Ageeva TS, Bukreeva EB, Khristoliubova EI. [Criteria and methods of etiological diagnosis of acute and chronic inflammatory processes in the lungs]. Ter Arkh. 1985;57(5):39-42. Russian. PMID 3895549
- [Background] Holte K, Kehlet H. Postoperative ileus: a preventable event. Br J Surg. 2000 Nov;87(11):1480-93. doi: 10.1046/j.1365-2168.2000.01595.x. PMID 11091234
- [Background] Choi H, Kim JH, Park JY, Ham BK, Shim Js, Bae JH. Gum chewing promotes bowel motility after a radical retropubic prostatectomy. Asia Pac J Clin Oncol. 2014 Mar;10(1):53-9. doi: 10.1111/ajco.12113. Epub 2013 Aug 12. PMID 23937408
- [Background] Li S, Liu Y, Peng Q, Xie L, Wang J, Qin X. Chewing gum reduces postoperative ileus following abdominal surgery: a meta-analysis of 17 randomized controlled trials. J Gastroenterol Hepatol. 2013 Jul;28(7):1122-32. doi: 10.1111/jgh.12206. PMID 23551339
- [Background] De Luca-Monasterios F, Chimenos-Kustner E, Lopez-Lopez J. [Effect of chewing gum on halitosis]. Med Clin (Barc). 2014 Jul 22;143(2):64-7. doi: 10.1016/j.medcli.2013.11.038. Epub 2014 Feb 20. Spanish. PMID 24559542
- [Background] Sasaki-Otomaru A, Sakuma Y, Mochizuki Y, Ishida S, Kanoya Y, Sato C. Effect of regular gum chewing on levels of anxiety, mood, and fatigue in healthy young adults. Clin Pract Epidemiol Ment Health. 2011;7:133-9. doi: 10.2174/1745017901107010133. Epub 2011 Aug 5. PMID 21866229
- [Background] Miles C, Johnson AJ. Chewing gum and context-dependent memory effects: a re-examination. Appetite. 2007 Mar;48(2):154-8. doi: 10.1016/j.appet.2006.07.082. Epub 2006 Oct 19. PMID 17055609
- [Background] Mickenautsch S, Leal SC, Yengopal V, Bezerra AC, Cruvinel V. Sugar-free chewing gum and dental caries: a systematic review. J Appl Oral Sci. 2007 Apr;15(2):83-8. doi: 10.1590/s1678-77572007000200002. PMID 19089107
- [Background] Zaghiyan K, Felder S, Ovsepyan G, Murrell Z, Sokol T, Moore B, Fleshner P. A prospective randomized controlled trial of sugared chewing gum on gastrointestinal recovery after major colorectal surgery in patients managed with early enteral feeding. Dis Colon Rectum. 2013 Mar;56(3):328-35. doi: 10.1097/DCR.0b013e31827e4971. PMID 23392147
- [Background] Cavusoglu YH, Azili MN, Karaman A, Aslan MK, Karaman I, Erdogan D, Tutun O. Does gum chewing reduce postoperative ileus after intestinal resection in children? A prospective randomized controlled trial. Eur J Pediatr Surg. 2009 Jun;19(3):171-3. doi: 10.1055/s-0029-1202776. Epub 2009 Apr 9. PMID 19360548
- [Background] Tamura T, Yatabe T, Kitagawa H, Yamashita K, Hanazaki K, Yokoyama M. Oral carbohydrate loading with 18% carbohydrate beverage alleviates insulin resistance. Asia Pac J Clin Nutr. 2013;22(1):48-53. doi: 10.6133/apjcn.2013.22.1.20. PMID 23353610